CLINICAL TRIAL: NCT04409405
Title: Evaluation and Support to Ebola Virus Disease Cured Patients and Their Contacts in the Democratic Republic of the Congo
Brief Title: Evaluation and Support to EVD Cured Patients and Their Contacts (Les Vainqueurs d'Ebola)
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-59; ESP/CE/287/2019 (Other: EC Kinshasa School of Public Health)
Record Dates: First submitted 2020-04-14; First posted 2020-06-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2022-02

CONDITIONS: Ebola Virus Disease
Keywords: Ebola; Democratic Republic of the Congo; DRC; Ituri; North Kivu
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample Urine Saliva Tear drop Breast milk Stool Vaginal fluid Semen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cured population: • Age ≥ 5 year old
- Contact population: * Age ≥ 5 year old
  * Contact of a participant included in cured-population cohort
  * Not diagnosed with EVD

SUMMARY:
Ebola virus is one of the most dangerous human pathogens and is an emerging public health problem in sub-Saharan Africa. Ebola virus disease (EVD) first appeared in 1976. The current epidemic in the Democratic Republic of the Congo (DRC) is one of the largest and most complex ever recorded, and is not yet under control: a new death has been reported on April 10th, 2020. The epidemic was declared a public health emergency of international scope by the World Health Organization (WHO) on July 17th, 2019.

Two studies are the "standard" in the assessment of the consequences of infection in survivors, in Liberia (PREVAIL) and Guinea (PostEbogui), especially in:

* The observation of comparable mortality rates, even if over time there was an improvement in survival, probably linked to the improvement in the quality of care and symptomatic treatment;
* And the study of the contacts of the survivors, between 4 to 10% of them had done seroconversion with regard to Ebola virus (EBOV) in an asymptomatic or pauci-symptomatic way and that this rate varied according to the degree of exposure to the risk.

The DRC's experience in this area and the enormous progress made in the fight against Viral hemorrhagic fevers (VHFs), therapeutically and preventively (where much of which patients have benefited from antiviral treatment or monoclonal antibodies), the technological responses (real-time sequencing of Ebola strains in new cases, vaccination or the use of individual isolation units), show the limits of their effectiveness. A large number of questions therefore remain unanswered:

* The antibody profile of the survivors, in particular the repertoire of immunoglobulin G (IgG) specific to these individuals and its correlation with survival and its evolution over time;
* The impact of treatments initiated during the acute phase on these immune abnormalities;
* Finally, genetic factors linked to the host could play an important role in the response to the Ebola virus.

The aim of this study is to provide a better overall understanding of Ebola virus infection and its clinical, virological, and immunological consequences, of cured people and their contacts; strengthen multidisciplinary monitoring of patients after an acute phase of EVD. The results will therefore have a direct impact on the clinical management of this population and on the prevention of possible secondary contamination in the Democratic Republic of the Congo.

ELIGIBILITY:
Inclusion Criteria:

In cured population

* Age ≥ 5 years
* Adults and children after an acute episode declared cured of biologically confirmed Ebola virus disease (two negative PCRs are required at least 24 hours apart so that a patient without clinical symptoms can leave the Ebola treatment center),
* Informed consent signed by at least one of the two parents or the legal guardian authorizing the child's participation in the study,
* Volunteer participant who signed the informed consent for adults.

In CONTACT population

* Age ≥ 5 years,
* Be a contact person of a cured patient (ie patient with a proven EVD, and with two negative PCRs at least 24 hours apart) included in the cohort of Ebola Winners. Based on WHO recommendations and the Centers for Disease Control and Prevention for the identification and traceability of contact subjects: a contact person is defined as a person who encountered the index case during his EVD in his residence, ie having the same place of life as him,
* Have not been diagnosed with EVD,
* Participation agreement:

  * For adult participants (≥ 18 years old, emancipated or married): informed consent intended for the adult participant signed,
  * For minors ≥ 5 years old: informed consent intended for the parent(s)/legal guardian signed by at least one of the two parents or the legal guardian and assent form intended for the minor participant completed.

In cellular immunological sub-study:

* Adult participants in the parent study ≥ 18 years old,
* Accept to participate in this sub-study
* Negative blood EBOV PCR

Exclusion Criteria:

* Absence of possible follow-up over 12 months from a logistical or geographical point of view (only for cured patients);
* Non-residents in the DRC;
* Impossibility of complying with the requirements and procedures of the study in the opinion of the investigator;
* Inability to consent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cured patients: study team will approach every declared-cured EBOV-infection patients discharged of a Ebola treatment center (Beni, Butembo, Mambassa or Mangina), older than 5 year old
  Contact participants: Cured participants will identify contact with who they were in contact when ill.
Sampling Method: Non-Probability Sample
Enrollment: 787 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Cured-participant population co-infections | Baseline (BL)
  Frequencies of co-infections (human immunodeficiency virus, hepatitis B virus, hepatitis C virus)
Cured-participant population co-morbidities at any time in the study | Baseline (BL), month 3, month 6, month 9, month 12, month 18
  Frequencies of co-morbidities including severity
Evolution over time of clinical consequences in cured participants | Baseline (BL), month 3, month 6, month 9, month 12, month 18
  Sequelae of EVD in cured participants and their evolution according to clinical characteristics and received treatment during hospitalisation.
Evolution over time of immunological consequences in cured participants | Baseline (BL), month 6, month 12
  Proportion and evolution of IgG subclasses against nucleoprotein, VP40 and glycoprotein from isolates Mayinga1976 and Kissidougou-Makona2014.
Evolution over time of virological consequences in cured participants | Baseline (BL), month 3, month 6, month 9, month 12, month 18
  Evolution of EBOV virus identified by polymerase chain reaction (PCR) in biological samples (blood, urine, feces, saliva, tears, breast milk (breastfeeding women), genital secretions (women aged 15 and over) and sperm (men aged 15 and over)).
Description of contact-participants Ebola-virus-exposure risk | Baseline (BL)
  Description of exposure to the confirmed index case (duration and repetition of exposure, possible protection used, state of contagiousness of the confirmed index case including clinical condition and viremia), prevalence of EVD (living or deceased, with whom the subject was in contact), vaccination status against EVD.
Asymptomatic or pauci-symptomatic Ebola infections in contact participants (clinical assessment) | Baseline (BL)
  Clinical assessment for EBOV infection since contact exposure to EVD patient.
Asymptomatic or pauci-symptomatic Ebola infections in contact participants (immunological assessment) | Baseline (BL)
  Titration of IgG subclasses against nucleoprotein, VP40 and glycoprotein.
Asymptomatic or pauci-symptomatic Ebola infections in contact participants (virological assessment) | Baseline (BL)
  Presence of Ebola virus identified by PCR in biological samples (blood, urine, feces, saliva, tears, breast milk (breastfeeding women), genital secretions and sperm (men aged 15 and over)).
Evolution over time of peripheral blood mononuclear cells (PBMC) in cured and contact participants (cellular immunological sub-study) | Baseline (BL), month 6, month 12
  Phenotypic characterization and activation status of the different cell populations within PBMC (T cells, B cells, natural killer cells, dendritic cells, etc.) by flow cytometry
Evolution over time of concentration of immune response analytes in cured and contact participants (cellular immunological sub-study) | Baseline (BL), month 6, month 12
  Titration of analytes involved in immune responses (using Luminex technology)
Evolution over time of EBOV-specific T responses in cured and contact participants (cellular immunological sub-study) | Baseline (BL), month 6, month 12
  EBOV-specific T responses after stimulation of cells by flow cytometry
Evolution over time of gene-expression profile in cured and contact participants (cellular immunological sub-study) | Baseline (BL), month 6, month 12
  Analysis of gene-expression profile in whole blood using Ilumina technology
Evolution over time of genetic heterogeneity in cured and contact participants (cellular immunological sub-study) | Baseline (BL), month 6, month 12
  Single-cell analysis to evaluate cellular genetic heterogeneity in cell population.
Genetic sub-study in cured and contact participants | Baseline (BL)
  Research of genetic variants implied in EBOV-infection response.

CONTACTS AND LOCATIONS:
Locations (4):
- Democratic Republic of the Congo (4):
  - Beni Hospital, Beni
  - Mangina Hospital, Beni
  - Butembo Hospital, Butembo
  - Mambasa Hospital, Mambasa

REFERENCES:
- [Background] Dilu-Keti A, Tovar-Sanchez T, Cuer B, Nkuba-Ndaye A, Mukadi-Bamuleka D, Panzi-Kalunda E, Kitenge-Omasumbu R, Bulabula-Penge J, Mambu-Mbika F, Mbala-Kingebeni P, Ayouba A, Muyembe-Tamfum JJ, Etard JF, Chenge F, Delaporte E, Ahuka-Mundeke S; 'Les Vainqueurs d'Ebola' study group. Long-term Sequelae in Ebola Virus Disease Survivors Receiving Anti-Ebola Virus Therapies in the Democratic Republic of the Congo: A Prospective Cohort Study. Open Forum Infect Dis. 2025 Jul 31;12(8):ofaf436. doi: 10.1093/ofid/ofaf436. eCollection 2025 Aug. PMID 40809394
- [Background] Nkuba-Ndaye A, Dilu-Keti A, Tovar-Sanchez T, Diallo MSK, Mukadi-Bamuleka D, Kitenge R, Formenty P, Legand A, Edidi-Atani F, Thaurignac G, Pelloquin R, Mbala-Kingebeni P, Toure A, Ayouba A, Muyembe-Tamfum JJ, Delaporte E, Peeters M, Ahuka-Mundeke S; Les Vainqueurs d'Ebola Study Group. Effect of anti-Ebola virus monoclonal antibodies on endogenous antibody production in survivors of Ebola virus disease in the Democratic Republic of the Congo: an observational cohort study. Lancet Infect Dis. 2024 Mar;24(3):266-274. doi: 10.1016/S1473-3099(23)00552-2. Epub 2023 Nov 30. PMID 38043556